CLINICAL TRIAL: NCT01806857
Title: The Experimental Treatment of Bulbar Dysfunction in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Clinical Trial Nuedexta in Subjects With ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Neurologic Study, La Jolla, California, (Other)
Collaborators: ALS Association (Other); State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Richard A. Smith, MD, Director, Center for Neurologic Study, La Jolla, California,
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2012P001274; 3FKVAD (Other Grant/Funding Number: ALSA)
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic lateral sclerosis; ALS; Nuedexta; Bulbar function; motor neurons
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — dextromethorphan - quinidine combination; Dextromethorphan; Quinidine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nuedexta then Matching Placebo (Other): Subjects in this arm will receive treatment with Nuedexta first for 28 days (±3 days) and then crossed over to receive treatment with matching placebo for 28 days (±3 days).
  Interventions: Drug: Nuedexta; Drug: Matching Placebo
- Matching Placebo then Nuedexta (Other): Subjects in this arm will receive treatment with matching placebo first for 28 days (±3 days) and then crossed over to receive treatment with Nuedexta for 28 days (±3 days).
  Interventions: Drug: Nuedexta; Drug: Matching Placebo

INTERVENTIONS:
Drug: Nuedexta — Nuedexta PO (by mouth) for 28 ± 3 days
  Other Names: dextromethorphan hydrobromide and quinidine sulfate
Drug: Matching Placebo — matching placebo PO (by mouth) for 28 ± 3 days
  Other Names: sugar pill

SUMMARY:
The purpose of this study is to determine whether Nuedexta is effective in the treatment of symptoms (impaired speech, swallowing, and saliva control)associated with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
Muscle weakness, the cardinal feature of ALS, leads to progressive loss of motor function affecting the limbs, tongue, respiratory and pharyngeal muscles. Symptomatic treatments such as the placement of a feeding tube, can compensate for the inability to swallow. Riluzole, the only approved treatment for ALS, may slow disease progression but no treatment is curative and none have improved function.

Unexpectedly, Nuedexta®, approved for the treatment of labile emotionality that occurs in association with ALS and other neurological disorders, has been observed to improve bulbar function, primarily speech and swallowing, in a number of neurological disorders, including ALS. The basis for this is conjectural but likely due to a direct effect of the drug on motor neurons in the part of the brain that controls speech and swallowing. The same part of the brain appears to modulate the expression of emotions and interestingly the site of action of the drug is the same as a site that has been implicated in a juvenile form of ALS.

This is a multicenter, randomized double-blind, placebo controlled, cross over study evaluating the palliative effect of Nuedexta® on bulbar dysfunction. It is expected that approximately 60 ALS patients from 7 clinical centers in the US will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria
* Age 18 years or older
* Exhibits bulbar dysfunction manifested by dysarthria and/or dysphagia, according to PI judgment, exhibits a score of 55 or above on the CNS-Bulbar Function Scale
* Capable of providing informed consent and following trial procedures
* Geographic accessibility to the site
* Women must not be able to become pregnant for the duration of the study and must be willing to be on two contraceptive therapies
* Slow vital capacity (SVC) measure ≥50% of predicted for gender, height, and age at the screening visit
* Must be able to swallow capsules throughout the course of the study, according to PI judgment
* Subjects must not have taken riluzole for at least 30 days or be on a 50mg BID dose of riluzole for at least 30 days prior to randomization (subjects how have never taken riluzole are permitted in the study)
* Subjects taking anti-sialorrhea medication(s) must be on a stable dose for at least 30 days prior to randomization (anti-sialorrhea naïve subjects are permitted in the study)
* Must be able to safely swallow at least 30 milliliters (mLs) of water for the water swallowing test

Exclusion Criteria:

* Prior use of Nuedexta®
* Current use of dextromethorphan, quinidine, quinine, mefloquine or opioids
* History of quinidine, quinine, or mefloquine-induced thrombocytopenia, hepatitis, or other hypersensitivity reactions
* History of known sensitivity or intolerability to dextromethorphan
* Use of an mono amine oxidase inhibitor (MAOI) or within 14 days of stopping an MAOI
* Prolonged QT interval, congenital long QT syndrome, history suggestive of torsades de pointes, or heart failure
* Complete atrioventricular (AV) block without implanted pacemaker, or subjects at high risk of complete AV block
* Concomitant use with drugs that both prolong QT interval and are metabolized by cytochrome P 2D6 (CYP2D6) (i.e., thioridazine or pimozide)
* Exposure to any other experimental agent (off-label use or investigational) within 30 days prior to Baseline Visit
* Invasive ventilator dependence, such as tracheostomy
* Any history of either substance abuse within the past year, unstable psychiatric disease, cognitive impairment, or dementia, according to PI judgment
* Placement and/or usage of feeding tube
* Pregnant women or women currently breastfeeding
* Unable to turn diaphragm pacing device off during swallowing tests
* Salivatory Botox within 90 days (3 months) of screening
* Salivatory radiation within 180 days (6 months) of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Smith, MD, Principal Investigator — Center for Neurologic Study (CNS); Jeremy Shefner, MD, PhD, Principal Investigator — Barrow Neurological Institute; Merit E Cudkowicz, MD, MSc, Principal Investigator — Massachusetts General Hospital (MGH)
Locations (7):
- United States (7):
  - California Pacific Medical Center, San Francisco, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Neurology Associates, P.C., Lincoln, Nebraska
  - The Cleveland Clinic, Cleveland, Ohio
  - Providence ALS Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Northeast ALS Consortium Website — http://www.alsconsortium.org/
- See also: ALS Association Website — http://www.alsa.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 90 subjects were consented for this trial, however, of the 90 that consented, 30 subjects were found to not meet eligibility criteria, and therefore were not treated.
Period: Overall Study
Arm/Group | Nuedexta Then Matching Placebo | Matching Placebo Then Nuedexta
Started | 31 | 29
Completed | 30 | 29
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients who signed a consent form and had a baseline visit.
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 58 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 34
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0
  Asian | 1
  Black/African American | 2
  Caucasian/White | 57
Region of Enrollment [Number; unit: participants]
  United States | 60
Baseline CNS-BFS Total Score [Mean (Standard Deviation); unit: units on a scale] — The Center for Neurologic Study-Bulbar Function Scale (CNS-BFS) is a 21-item self report scale that assesses three domains of bulbar function: speech, swallowing and salivation (sialorrhea). Scores for each question range from 1 (does not apply) to 5 (applies most of the time). The higher the score, the worse the speech, swallowing and salivation (sialorrhea). [Range of score: 21-105]
  units on a scale | 58.15 (13.37)
Baseline ALSFRS-R Total Score [Mean (Standard Deviation); unit: units on a scale] — The ALSFRS-R is a quickly administered (5 min) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
  units on a scale | 34.58 (6.95)
Baseline CNS Lability Scale Total Score [Mean (Standard Deviation); unit: units on a scale] — The Center for Neurologic Study-Lability Scale (CNS-LS) is a 7-item self report scale that assesses pseudobulbar affect (PBA) by measuring the perceived frequency of PBA episodes (laughing or crying). Each item is scored using a 5-point Likert scale, from 1 (applies never) to 5 (applies most of the time). Scores range from 5-35.
  units on a scale | 13.67 (5.55)

OUTCOME MEASURES:

1. Primary Outcome: Bulbar Function Scale (CNS-BFS) Total Score
Description: The Center for Neurologic Study-Bulbar Function Scale (CNS-BFS) is a 21-item self report scale that assesses three domains of bulbar function: speech, swallowing and salivation. Scores for each question range from 1 (does not apply) to 5 (applies most of the time). The higher the score, the worse the speech, swallowing and salivation (sialorrhea). [Range of score: 21-105]
  The scale was modeled on the Center for Neurologic Study Emotional Lability Scale (CNS-LS) that has been a robust endpoint in four clinical trials. The scale was validated in a large population of ALS patients (n=122) and detects impaired bulbar function at a sensitivity of 90% and a specificity of 0.97%. Test re-test correlation was 0.92% at six-months (n=53).
Time Frame: Average between Screening Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Neudexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 53.45 (1.07) | 59.31 (1.1)
Statistical Analysis 1: Comparison: Active Drug (Neudexta) vs Matching Placebo; Test type: Superiority or Other; p = 0.0003, Random Effects Model

2. Primary Outcome: Bulbar Function Scale (CNS-BFS) Sialorrhea Score
Description: The Center for Neurologic Study-Bulbar Function Scale (CNS-BFS) is a 21-item self report scale that assesses three domains of bulbar function: speech, swallowing and salivation. Scores for each question range from 1 (does not apply) to 5 (applies most of the time). The higher the score, the worse the salivation (sialorrhea). There are 7 salivation (sialorrhea) questions, with a score range of 7 to 35.
Time Frame: Average between Screening Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Neudexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 14.28 (0.37) | 15.81 (0.38)

3. Primary Outcome: Bulbar Function Scale (CNS-BFS) Speech Score
Description: The Center for Neurologic Study-Bulbar Function Scale (CNS-BFS) is a 21-item self report scale that assesses three domains of bulbar function: speech, swallowing and salivation. Scores for each question range from 1 (does not apply) to 5 (applies most of the time). The higher the score, the worse the speech. There are 7 speech questions, with a score range of 7 to 35.
Time Frame: Average between Screening Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Neudexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 22.22 (0.56) | 24.57 (0.57)

4. Primary Outcome: Bulbar Function Scale (CNS-BFS) Swallowing Score
Description: The Center for Neurologic Study-Bulbar Function Scale (CNS-BFS) is a 21-item self report scale that assesses three domains of bulbar function: speech, swallowing and salivation. Scores for each question range from 1 (does not apply) to 5 (applies most of the time). The higher the score, the worse the swallowing. There are 7 swallowing questions, with a score range of 7 to 35.
Time Frame: Average between Screening Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Neudexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 17.14 (0.46) | 18.92 (0.47)

5. Secondary Outcome: Center for Neurologic Study - Lability Scale (CNS-LS) Total Score
Description: The Center for Neurologic Study-Lability Scale (CNS-LS) is a 7-item self report scale that assesses pseudobulbar affect (PBA) by measuring the perceived frequency of PBA episodes (laughing or crying). Each item is scored using a 5-point Likert scale, from 1 (applies never) to 5 (applies most of the time). Scores range from 5-35. The higher the score, the worse the PBA.
Time Frame: Average between Screening Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 10.79 (0.47) | 13.72 (0.49)
Statistical Analysis 1: Comparison: Active Drug (Nuedexta) vs Matching Placebo; Test type: Superiority or Other; p = 0.0001, Random Effects Model

6. Secondary Outcome: ALS Functional Rating Scale- Revised (ALSFRS-R) Total Score
Description: The ALSFRS-R is a quickly administered (5 min) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
Time Frame: Average between Screening Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 34.15 (0.33) | 33.7 (0.33)

7. Secondary Outcome: Visual Analog Scale - Speech Scores
Description: Visual analog scales are useful for measuring complex clinical events and offer the advantage of self-administration and responsiveness to change over time. The scales designed for this study inventory three domains of bulbar function: speech, swallowing and salivation (sialorrhea). For each of these, subjects score themselves by indicating their level of function on a scale of 1 (severe impairment) to 10 (normal). Scores range from 1 to 10; the higher the score, the more normal the function.
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 4.97 (0.21) | 4.11 (0.21)

8. Secondary Outcome: Ashworth Spasticity Scale Score - Right Arm
Description: This is a standard measure for spasticity that has been used in numerous ALS clinical trials to assess spasticity due to upper motor neuron dysfunction in ALS. Data is generated from the clinical exam and scored from 1-5, the lowest score indicating normal tone and the highest muscle rigidity.
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 1.65 (0.06) | 1.53 (0.06)

9. Secondary Outcome: Timed Reading of Test Paragraph Result
Description: Subjects will be asked to read 'The Rainbow Passage' a commonly used test paragraph utilized by speech pathologists to assess speech rate (words/minute). Study staff will time the subject to determine how many words the subject reads per minute. It is used primarily because it contains every sound in the English language. Subjects will also be observed for loudness, nasality, and intelligibility.
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: words per minute
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
words per minute | 107.12 (1.79) | 103.37 (1.83)

10. Secondary Outcome: Average Water Swallowing Test (WST)
Description: The Water Swallowing Test (WST) estimates swallowing speed, a useful and reproducible measure. While sitting, subjects are asked to drink 30 milliliters (mL) of liquid. The time for subjects to complete this task is a sensitive measure for the detection of swallowing dysfunction and is a simple measure for serial assessment of subjects. The test will be completed three times, with the best two scores recorded to obtain an average score. Following completion of the WST, the subject's swallowing abilities (choking, spillage, and effort) will be observed.
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
seconds | 12.16 (0.71) | 13.11 (0.72)

11. Secondary Outcome: Visual Analog Scale - Swallowing Score
Description: as for outcome 7
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 7.23 (0.29) | 6.93 (0.3)

12. Secondary Outcome: Visual Analog Scale - Salivation (Sialorrhea) Score
Description: as for outcome 7
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 6.78 (0.31) | 6.78 (0.32)

13. Secondary Outcome: Average Solids Swallowing Test
Description: The Time Swallowing Test assesses the subject's ability to swallow solids. For this test, the subject will be asked to consume a tablespoon of cereal containing 5 cheerios. The subject will be instructed to close their mouth, chew and subsequently swallow the bolus. The time to complete this task will be recorded. The test will be completed three times to obtain an average score.
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
seconds | 18.53 (1.16) | 19.45 (1.19)

14. Secondary Outcome: Ashworth Spasticity Scale Score - Left Arm
Description: as for outcome 8
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 1.62 (0.06) | 1.67 (0.07)

15. Secondary Outcome: Ashworth Spasticity Scale Score - Right Leg
Description: as for outcome 8
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 1.94 (0.1) | 1.82 (0.1)

16. Secondary Outcome: Ashworth Spasticity Scale Score - Left Leg
Description: as for outcome 8
Time Frame: Average between Baseline Visit to Visit 3
Population: Includes all participants that received at least one dose of intervention.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Drug (Nuedexta) | Matching Placebo
Number analyzed (Participants) | 58 | 57
units on a scale | 1.91 (0.09) | 1.91 (0.09)

ADVERSE EVENTS:
Time Frame: 28 days +/- 3 days for each Intervention.
Description: Safety population included all participants who received at least one dose of intervention.
Groups:
- Active Drug (Neudexta): Includes all subjects that took the active drug (Neudexta)
- Matching Placebo: Includes all subjects that took matching placebo
Arm/Group | Active Drug (Neudexta) | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/57
Other Adverse Events (participants affected / at risk) | 21/58 | 4/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug (Neudexta) (N=58) | Matching Placebo (N=57)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug (Neudexta) (N=58) | Matching Placebo (N=57)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Dizziness (Nervous system disorders) | 7 (10) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes